CLINICAL TRIAL: NCT04441905
Title: A Phase 1, Randomized, Double-Blind, Multi-Site, Single Dose Escalation Study to Evaluate the Safety, Pharmacokinetics, and Immunogenicity of SAR440894 vs Placebo in Healthy Adults
Brief Title: Phase 1 Study of SAR440894 vs Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-0006
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09-11

CONDITIONS: Chikungunya Virus Infection
Keywords: Chikungunya Virus; dose escalation; healthy adults; Immunogenicity; Pharmacokinetics; phase 1; placebo; SAR440894
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 (Experimental): 0.3 mg/kg of SAR440894 (n=6) or placebo (n=2) administered once during a 60-minute intravenous (IV) infusion. 2 sentinel subjects will receive dosing for review of safety data (SAR440894 n=1, placebo n=1) before remainder of cohort.
  Interventions: Other: Placebo; Biological: SAR440894
- Cohort 2 (Experimental): 1 mg/kg of SAR440894 (n=6) or placebo (n=2) administered once during a 60-minute intravenous (IV) infusion. 2 sentinel subjects will receive dosing for review of safety data (SAR440894 n=1, placebo n=1) before remainder of cohort.
  Interventions: Other: Placebo; Biological: SAR440894
- Cohort 3 (Experimental): 3 mg/kg of SAR440894 (n=6) or placebo (n=2) administered once during a 60-minute intravenous (IV) infusion. 2 sentinel subjects will receive dosing for review of safety data (SAR440894 n=1, placebo n=1) before remainder of cohort.
  Interventions: Other: Placebo; Biological: SAR440894
- Cohort 4 (Experimental): 10 mg/kg of SAR440894 (n=6) or placebo (n=2) administered once during a 60-minute intravenous (IV) infusion. 2 sentinel subjects will receive dosing for review of safety data (SAR440894 n=1, placebo n=1) before remainder of cohort.
  Interventions: Other: Placebo; Biological: SAR440894
- Cohort 5 (Experimental): 20 mg/kg of SAR440894 (n=6) or placebo (n=2) administered once during a 60-minute intravenous (IV) infusion. 2 sentinel subjects will receive dosing for review of safety data (SAR440894 n=1, placebo n=1) before remainder of cohort.
  Interventions: Other: Placebo; Biological: SAR440894

INTERVENTIONS:
Other: Placebo — One time 60-minute IV infusion of lyophilized placebo for SAR440894
Biological: SAR440894 — One time 60-minute IV infusion of SAR440894 monoclonal antibody (IgG1) directed against the E2 envelope protein of chikungunya virus

SUMMARY:
A single, ascending-dose design with five dose-cohorts of 8 subjects. Forty healthy adults aged 18 to 45, inclusive, will be recruited and admitted at multiple sites. Each subject will be randomized to receive either SAR440894 or matching placebo via 60-minute intravenous infusion. In each cohort of 8 subjects, the randomization ratio will be 6 active to 2 placebo, and 2 sentinel subjects (one from each active and placebo group) will be dosed first. Dosing of the next dose-cohort will be dependent on acceptable meeting predefined safety criteria in the preceding cohort. Each subject's participation will take place over approximately 150 days, not including the screening visit. There are no hypotheses for this phase I study. The primary objective will be to determine the safety of single ascending intravenous (IV) infusions of SAR440894 when administered in healthy adults.

DETAILED DESCRIPTION:
A single, ascending-dose design with five dose-cohorts of 8 subjects. Forty healthy adults aged 18 to 45, inclusive, will be recruited and admitted at multiple sites. Each subject will be randomized to receive either SAR440894 or matching placebo via 60-minute intravenous infusion. In each cohort of 8 subjects, the randomization ratio will be 6 active to 2 placebo, and 2 sentinel subjects (one from each active and placebo group) will be dosed first. Dosing of the next dose-cohort will be dependent on acceptable meeting predefined safety criteria in the preceding cohort. Each subject's participation will take place over approximately 150 days, not including the screening visit. There are no hypotheses for this phase I study. The primary objective will be to determine the safety of single ascending intravenous (IV) infusions of SAR440894 when administered in healthy adults. The secondary objectives are: 1) to determine the pharmacokinetics (PK) of single ascending doses of 60-minute IV infusions SAR440894 in healthy adults and 2) to asses the immunogenicity of single ascending doses of 60-minute IV infusions SAR440894 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a healthy adult 18 to 45 years of age, inclusive, with a body mass index (BMI) greater than 18 or less than 35 kg/m^2, inclusive.
2. Participants of childbearing potential* having vaginal intercourse must use an effective method of contraception** from 45 days before study product administration through the final study visit.

   *Not sterilized via hysterectomy or bilateral oophorectomy and/or salpingectomy or be less than 1 year from the last menses if menopausal.

   **Includes any of the following (a) exclusive non-male sexual relationships; (b) monogamous relationship with vasectomized partner (greater than or equal to 180 days between procedure and subject receipt of investigational product); (c) bilateral tubal ligation or tubal occlusion (eg., Essure(R)); (d) effective intrauterine device (IUD); (e) hormonal implants (eg., Implanon(R)); (f) other hormonal contraceptives (such as birth control pills, vaginal rings, patches or injections); (g) barrier methods (condom, diaphragm, cervical cap) PLUS spermicide (gel or foam)
3. Women of childbearing potential must agree not to donate ova or oocytes (ie, human eggs) during the study.
4. Male subjects (including those with vasectomies) whose partners are of childbearing potential should use condoms with spermicide and not donate sperm for the duration of the study.
5. Must have adequate venous access for IV infusions and blood draws.
6. Agrees to be available for all study visits and willing to cooperate fully with the requirements* of the study protocol.

   *Requirements include remaining in confinement for at least 72 hours after receiving study product and other activities outlined in the protocol's Schedule of Events.
7. Is able to understand the informed consent process and procedures and signs the consent form.
8. Will agree not to donate any blood or blood products* for the duration of the study.

   * Includes whole blood, red blood cells, platelets, plasma, or plasma derivatives.
9. Will agree to avoid travel to endemic areas (as defined by the Center for Disease Control (CDC)) for Chikungunya Virus (CHIKV) at any point during the Follow-up period (https://www.cdc.gov/chikungunya/geo/index.html).

Exclusion Criteria:

1. Has any medical condition (renal dysfunction) that, in the opinion of the site PI or appropriate sub-investigator listed on Form Food and Drug Administration (FDA) 1572, is a contraindication to study participation.
2. Has any clinically significant (CS) electrocardiogram (ECG) abnormalities in the opinion of the site Principal Investigator (PI) or appropriate sub-investigator been listed on Form FDA 1572.
3. Use of any prohibited prescription medication (excluding contraceptives in females) within 14 days before study product administration, through Day 56** *Prohibited medications include immunosuppressives; immune modulators; oral corticosteroids (topical/intranasal steroids are acceptable); prescription Non-Steroidal Anti-inflammatory Drugs (NSAIDs); anti-neoplastic agents; any vaccine (licensed or investigational). If study activities overlap with the influenza season, subjects will be instructed to obtain influenza vaccine at least 45 days prior to proposed dosing or delay vaccination until after Day 56. Subjects will be instructed to obtain the last dose of any vaccine for SARS-CoV-2 (COVID-19) at least 45 days prior to proposed dosing or delay vaccination until after Day 56.
4. Use of nonprescription systemic drugs within 7 days before study product administration (includes vitamins, antacids*, over-the-counter drugs**, herbal/dietary supplements, etc.) through Day 28***

   *Nonprescription drugs and supplements may be allowed before Day 28 at the discretion of the site PI.

   **Includes proton pump inhibitors and H2-blockers (Histamine-2 blockers)

   ***Nonprescription drugs and supplements may be allowed before Day 28 at the discretion of the site PI. In the event an OTC oral contraceptive becomes available during the course of the study, it must be reviewed and approved by the site PI.
5. Hypertension, with confirmed systolic blood pressure (BP) greater than 140 mm Hg or confirmed diastolic BP greater than 90 mm Hg, measured after 5 minutes of rest at Screening.
6. Hypotension, with confirmed systolic BP less than 90 mm Hg.
7. Resting heart rate (HR) less than 45 bpm or greater than 100 bpm at Screening.
8. Body weight less than 50 kg.
9. History of a significant illness, per the investigators' clinical judgment, within 2 weeks before dosing (subjects can screen after illness is resolved for 2 weeks).
10. Known diagnosis of prolonged QT interval, congenital long QT syndrome, bradyarrhythmias, or uncompensated heart failure.
11. Males with a mean QTcF greater than 450 msec or females with a mean QTcF greater than 470 msec (Fridericia's correction) at Screening.*

    *ECG tracings should be recorded at least 1 minute apart, after at least 5 minutes of rest in the supine position. If the mean QTcF value from the 3 tracings exceeds the limits stated, the subject is disqualified.
12. Any history of malignancy ever, except low-grade skin cancer (ie, basal cell carcinoma thought to be cured).
13. History of drug abuse, alcohol abuse, or significant psychiatric history according to the investigators' judgment within 12 months before Screening.
14. Positive for hepatitis B virus surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody at Screening.
15. Excessive consumption of beverages containing xanthine bases, or more than 400 mg of caffeine per day within 1 week of study product administration through the final study visit.
16. Consumption of alcohol within 24 hours before study product administration.
17. Use of nicotine-containing products within 45 days before study product administration through the final study visit.
18. Positive drug screen*, positive cotinine screen, or positive breathalyzer test for alcohol at Screening or admission (Day -1).

    *Cannabinoids, amphetamines, barbiturates, cocaine, opiates, benzodiazepines and phencyclidine. Subjects should be notified by phone not to consume any poppy seeds within 24 hours before the Screening urine test to avoid a false positive opioid test result.
19. If female, serum positive pregnancy test at Screening or serum positive pregnancy test on Day -1.
20. Breastfeeding throughout the duration of the study
21. Total WBC and platelet counts, hemoglobin*, total bilirubin*, alanine/aspartate aminotransferase* and sodium* are Grade 1 or higher** at Screening visit***.

    *For sodium; potential subjects excluded prior to Protocol Version 6.0 with Grade 1 sodium values may be rescreened.

    For hemoglobin; a lower limit within 0.5 g/dL of the lower limit of normal (LLN) is allowable at Screening.

    For total bilirubin; ULN values will be allowed at Screening and Day -1/baseline provided the AST and ALT are within normal limits. Potential subjects excluded prior to Protocol Version 6.0 with bilirubin values below the Version 6.0 upper limit may be rescreened.
    * For ALT/AST; subjects who screened prior to Protocol Version 11.0 were excluded if AST/ALT results were Grade 1 or higher at Screening. Subjects who screen with Protocol Version 11.0, AST/ALT is exclusionary if Screening results are 1.5 × ULN or if assessed as CS by the site PI.
    * Grade 1 or higher toxicity, see Appendix C and Appendix D for subjects who screened and enrolled prior to Protocol Version 11.0. Subjects who screen and enroll with Protocol Version 11.0, toxicity will be assessed with the NCI CTCAE, Version 5.0 - November 2017. Safety laboratory tests drawn on Day -1 or Screening if within 48 hours of planned dosing will serve as baseline values. Day -1 laboratory tests with a Grade 1 severity, other than those noted above, will not exclude subjects from participation.

      * All other abnormal laboratory values collected at Screening and on Day -1 will be exclusionary at the discretion of the PI.
22. Potassium, bicarbonate or creatinine/eGFR* results are Grade 1 or higher at either Screening or Day -1/Baseline visits.

    *For creatinine; subjects who screened prior to Protocol Version 11.0 were excluded if creatinine results were Grade 1 or higher. Subjects who screen with Protocol Version 11.0, creatinine is not an exclusionary criterion, instead subjects should have a calculated eGFR using Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation (CKD-EPI) of >/= 90 mL/min/1.73m2 to be enrolled in the study.
23. Received an experimental agent (vaccine, drug, biologic, device, or medication) within 45 days or 5 half-lives (whichever is longer) before study product administration.*

    *Prior participation at any time in noninvasive methodology trials in which no drugs were given is acceptable.
24. Is participating in or plans to participate in another clinical trial with an interventional agent that will be received during this trial.
25. Has donated more than 500 mL of blood or blood products* within the month before Screening.

    *Includes whole blood, red blood cells, platelets, plasma, or plasma derivatives.
26. Has a history of serologically-proven Chikungunya virus (CHIKV) exposure at any point, or positive anti CHIKV antibodies (ie., positive IgM or IgG) at Screening.
27. Has received blood products within 120 days prior to Screening.
28. Has received mAb in the past 3-months or 5 half-lives (whichever is longer) prior to Screening, whether licensed or investigational, or plans to receive a mAb outside of this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pharmaceutical Product Development - Orlando Clinical Research Unit, Orlando, Florida
  - Duke University School of Medicine - Duke Clinical Research Institute - Duke Clinical Research Unit, Durham, North Carolina
  - PPD - Austin Clinical Research Unit, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included healthy male and female adults, ages 18-45, inclusive, who met all eligibility criteria. Participants were enrolled at three sites in the United States between December 14, 2020 and March 25, 2024 and were recruited via IRB-approved procedure and materials, such as a participant-recruitment database, websites, outreach events, and electronic or other media.
Groups:
- Cohort 1 - SAR440894 0.3 mg/kg: 0.3 mg/kg of SAR440894 administered once during a 60-minute intravenous (IV) infusion.
  SAR440894: One time 60-minute IV infusion of SAR440894 monoclonal antibody (IgG1) directed against the E2 envelope protein of chikungunya virus
- Cohort 2 - SAR440894 1 mg/kg: 1 mg/kg of SAR440894 administered once during a 60-minute intravenous (IV) infusion.
  SAR440894: One time 60-minute IV infusion of SAR440894 monoclonal antibody (IgG1) directed against the E2 envelope protein of chikungunya virus
- Cohort 3 - SAR440894 3 mg/kg: 3 mg/kg of SAR440894 administered once during a 60-minute intravenous (IV) infusion.
  SAR440894: One time 60-minute IV infusion of SAR440894 monoclonal antibody (IgG1) directed against the E2 envelope protein of chikungunya virus
- Cohort 4 - SAR440894 10 mg/kg: 10 mg/kg of SAR440894 administered once during a 60-minute intravenous (IV) infusion.
  SAR440894: One time 60-minute IV infusion of SAR440894 monoclonal antibody (IgG1) directed against the E2 envelope protein of chikungunya virus
- Cohort 5 - SAR440894 20 mg/kg: 20 mg/kg of SAR440894 administered once during a 60-minute intravenous (IV) infusion.
  SAR440894: One time 60-minute IV infusion of SAR440894 monoclonal antibody (IgG1) directed against the E2 envelope protein of chikungunya virus
- Placebo: Placebo participants from Cohorts 1, 2, 3, 4, and 5. Placebo was administered by the same route as active drug.
  Placebo: One time 60-minute IV infusion of lyophilized placebo for SAR440894
Period: Overall Study
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Started | 6 | 7 | 6 | 6 | 7 | 10
Completed | 5 | 6 | 6 | 6 | 6 | 10
Not Completed | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Enrolled but treatment not administered | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Became ineligible after enrollment | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 7 | 10 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (7.9) | 39.0 (5.3) | 36.0 (8.9) | 37.2 (5.2) | 31.6 (7.2) | 28.9 (8.0) | 33.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 4 | 3 | 5 | 23
  Male | 3 | 3 | 2 | 2 | 4 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 5 | 0 | 5 | 5 | 18
  Not Hispanic or Latino | 5 | 5 | 1 | 6 | 2 | 5 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 3 | 3 | 3 | 15
  White | 2 | 4 | 5 | 3 | 4 | 7 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.12 (4.42) | 29.67 (4.91) | 27.95 (4.41) | 29.53 (3.45) | 26.94 (3.66) | 26.71 (2.52) | 27.74 (3.87)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events (AEs)
Description: The number of participants who experienced at least one unsolicited AE. An AE is defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product. Any medical condition that was present at screening was considered a baseline finding and not reported as an AE. However, if the severity (i.e., grade) of any pre-existing medical condition increases, it was recorded as an AE. For participants who enrolled prior to protocol v11.0, AEs were assessed with protocol defined criteria. For participants who enrolled under protocol v11.0, AEs were assessed with NCI CTCAE, Version 5.0.
Time Frame: Day 1 through Day 150
Population: The safety population includes participants who receive any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants | 5 | 3 | 2 | 3 | 2 | 6

2. Primary Outcome: Frequency of Serious Adverse Events (SAEs)
Description: The number of participants who experienced at least one SAE throughout the course of the study. An AE is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes:
  * Death
  * A life-threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
  * A congenital anomaly/birth defect.
Time Frame: Day 1 through Day 150
Population: The safety population includes participants who receive any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Frequency of Clinically Significant Vital Signs Results
Description: The number of participants who experienced at least one clinically significant vital signs abnormality post-dosing is summarized by parameter. Clinical significance was determined by the site investigator for all results that met toxicity grading criteria. For participants who enrolled prior to protocol v11.0, vital signs results were graded according to protocol-defined toxicity criteria. For participant who enrolled under protocol v11.0, vital signs results were graded according to the NCI CTCAE, Version 5.0.
Time Frame: Day 1 through Day 150
Population: The safety population includes participants who receive any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Systolic Blood Pressure (High) | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure (Low) | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure | 0 | 0 | 0 | 0 | 0 | 0
  Heart Rate (High) | 0 | 0 | 0 | 0 | 0 | 0
  Heart Rate (Low) | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Rate | 0 | 0 | 0 | 0 | 0 | 0
  Temperature | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Frequency of Clinically Significant Chemistry Laboratory Results
Description: The number of participants who experienced at least one clinically significant chemistry laboratory abnormality post-dosing is summarized by parameter. Clinical significance was determined by the site investigator for all results that were outside the normal range. For participants who enrolled prior to protocol v11.0, laboratory results were graded according to protocol-defined toxicity criteria. For participants who enrolled under protocol v11.0, laboratory results were graded according to the NCI CTCAE, Version 5.0.
Time Frame: Day 1 through Day 150
Population: The safety population includes participants who receive any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Sodium (Low) | 0 | 0 | 0 | 0 | 0 | 0
  Sodium (High) | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (Low) | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (High) | 0 | 0 | 0 | 0 | 0 | 0
  Bicarbonate (Low) | 0 | 0 | 0 | 0 | 0 | 0
  Bicarbonate (High) | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (Low) | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (High) | 0 | 1 | 0 | 0 | 0 | 1
  Blood Urea Nitrogen | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine | 0 | 0 | 0 | 0 | 0 | 0
  eGFR | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (Low) | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (High) | 0 | 0 | 0 | 0 | 0 | 0
  Albumin | 0 | 0 | 0 | 0 | 0 | 1
  Total Protein | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase | 0 | 0 | 0 | 0 | 0 | 0
  AST | 0 | 0 | 0 | 0 | 0 | 0
  ALT | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin | 0 | 0 | 0 | 0 | 0 | 0
  Cystatin-C | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Frequency of Clinically Significant Hematology Laboratory Results
Description: The number of participants who experienced at least one clinically significant hematology laboratory abnormality post-dosing is summarized by parameter. Clinical significance was determined by the site investigator for all results that were outside the normal range. For participants who enrolled prior to protocol v11.0, laboratory results were graded according to protocol-defined toxicity criteria. For participants who enrolled under protocol v11.0, laboratory results were graded according to the NCI CTCAE, Version 5.0.
Time Frame: Day 1 through Day 150
Population: The safety population includes participants who receive any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Hemoglobin (Low) | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (High) | 0 | 0 | 0 | 0 | 0 | 0
  WBC (Low) | 0 | 0 | 0 | 0 | 0 | 0
  WBC (High) | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (Low) | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (High) | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils | 0 | 0 | 0 | 0 | 1 | 0
  Eosinophils | 0 | 0 | 0 | 0 | 0 | 0
  Platelets | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit | 0 | 0 | 0 | 0 | 0 | 0
  RBC | 0 | 0 | 0 | 0 | 0 | 0
  Basophils | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Frequency of Clinically Significant Coagulation Laboratory Results
Description: The number of participants who experienced at least one clinically significant coagulation laboratory abnormality post-dosing is summarized by parameter. Clinical significance was determined by the site investigator for all results that were outside the normal range. For participants who enrolled prior to protocol v11.0, laboratory results were graded according to protocol-defined toxicity criteria. For participants who enrolled under protocol v11.0, laboratory results were graded according to the NCI CTCAE, Version 5.0.
Time Frame: Day 1 through Day 150
Population: The safety population includes participants who receive any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Activated Partial Thromboplastin Time | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin Time | 0 | 0 | 0 | 0 | 0 | 0
  INR | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Frequency of Clinically Significant Urinalysis Laboratory Results
Description: The number of participants who experienced at least one clinically significant urinalysis laboratory abnormality post-dosing is summarized by parameter. Clinical significance was determined by the site investigator for all results that were outside the normal range. For participants who enrolled prior to protocol v11.0, laboratory results were graded according to protocol-defined toxicity criteria. For participants who enrolled under protocol v11.0, laboratory results were graded according to the NCI CTCAE, Version 5.0.
Time Frame: Day 1 through Day 150
Population: The safety population includes participants who receive any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Urine Protein | 0 | 0 | 0 | 0 | 0 | 0
  Urine Glucose | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite | 0 | 0 | 0 | 0 | 0 | 0
  Occult Blood | 0 | 0 | 0 | 0 | 0 | 0
  Urine WBC | 0 | 0 | 0 | 1 | 1 | 0
  Urine RBC | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen | 0 | 0 | 0 | 0 | 0 | 0
  Ketones | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte Esterase | 0 | 0 | 0 | 1 | 0 | 0

8. Primary Outcome: Frequency of Clinically Significant Electrocardiogram (ECG) Results
Description: The number of participants who experienced at least one clinically significant ECG result post-dosing. Clinical significance was determined by the site investigator.
Time Frame: Day 1 through Day 150
Population: The safety population includes participants who receive any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Maximum Concentration (Cmax) of SAR440894 in Plasma
Description: PK parameters were estimated from the SAR440894 plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis.
Time Frame: Day 1 through Day 150
Population: The PK Population includes all participants who received a complete dose of SAR440894 and have at least one quantifiable post-dose plasma drug concentration record.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ug/mL | 7.2444 (34) | 29.1216 (25) | 91.8476 (8) | 307.1714 (16) | 466.6280 (14)

10. Secondary Outcome: Minimum Concentration (Cmin) of SAR440894 in Plasma
Description: as for outcome 9
Time Frame: Day 1 through Day 150
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ug/mL | 1.1677 (59) | 2.9886 (20) | 5.1829 (284) | 35.3937 (33) | 59.7625 (63)

11. Secondary Outcome: Time of Maximum Concentration (Tmax) of SAR440894 in Plasma
Description: as for outcome 9
Time Frame: Day 1 through Day 150
Population: as for outcome 9
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h | 2.10 [1.0 to 49] | 2.05 [1.0 to 2.3] | 5.00 [1.0 to 9.3] | 3.65 [1.0 to 9.0] | 2.00 [1.0 to 2.1]

12. Secondary Outcome: Time of Minimum Concentration (Tmin) of SAR440894 in Plasma
Description: as for outcome 9
Time Frame: Day 1 through Day 150
Population: as for outcome 9
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h | 3097.0 [342 to 3576] | 3542.5 [1993 to 3578] | 3578.0 [2666 to 3578] | 3530.5 [3338 to 3676] | 3577.0 [3485 to 3629]

13. Secondary Outcome: Area Under the Concentration-Time Curve From 0 h (Pre-Dose) to the Lase Concentration Above the Lower Limit of Quantitation (AUC0-last) of SAR440894 in Plasma
Description: as for outcome 9
Time Frame: Day 1 through Day 150
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ug*h/mL | 5108.6 (76) | 24191.0 (11) | 68548.3 (27) | 268599.9 (23) | 437019.3 (25)

14. Secondary Outcome: Area Under the Concentration-Time Curve From 0 h (Pre-Dose) to Infinity (AUC0-inf) of SAR440894 in Plasma
Description: PK parameters were estimated from the SAR440894 plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. AUC0-inf was estimated for parameters meeting the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) >= 0.90 and includes at least 3 time points after Tmax.
Time Frame: Day 1 through Day 150
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6
ug*h/mL | 9083.8 (19) | 30661.2 (11) | 85239.6 (44) | 364777.5 (27) | 693676.5 (55)

15. Secondary Outcome: Terminal Phase Elimination Rate Constant (Lambda-z) of SAR440894 in Plasma
Description: as for outcome 14
Time Frame: Day 1 through Day 150
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6
1/h | 0.0004111 (19) | 0.0004631 (17) | 0.0005153 (87) | 0.0003884 (30) | 0.0002922 (68)

16. Secondary Outcome: Terminal Half-Life (t1/2) of SAR440894 in Plasma
Description: as for outcome 14
Time Frame: Day 1 through Day 150
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6
h | 1687.0 (19) | 1497.9 (17) | 1344.0 (87) | 1784.0 (30) | 2373.0 (68)

17. Secondary Outcome: Clearance (CL) of SAR440894 in Plasma
Description: as for outcome 14
Time Frame: Day 1 through Day 150
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6
mL/h/kg | 0.0331 (19) | 0.0328 (11) | 0.0352 (44) | 0.0275 (27) | 0.0288 (55)

18. Secondary Outcome: Volume of Distribution (Vd) of SAR440894 in Plasma
Description: as for outcome 14
Time Frame: Day 1 through Day 150
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6
mL/kg | 80.38 (29) | 70.47 (20) | 68.25 (39) | 70.55 (34) | 98.72 (18)

19. Secondary Outcome: Incidence of Anti-drug Antibody (ADA) Assay Results
Description: Incidence of ADA is defined as either treatment-induced or treatment-boosted ADA at any time point post dosing. For immunogenicity assays, a positive result is defined as a positive screening assay followed by a positive confirmation assay. Treatment-induced ADA is defined as a negative result at baseline and a positive result post-dose. Treatment-boosted ADA is defined as a positive result at both baseline and post-dose, with a 4-fold increase in titer.
Time Frame: Day 1 through Day 150
Population: The Immunogenicity Population includes all participants who receive any amount of study product and contribute at least one post-infusion plasma sample for immunogenicity testing for which valid results are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs were documented from time of drug administration (Day 1) through the time of the last assessment (Day 150).
Description: For participants who enrolled prior to protocol v11.0, AEs were graded according to protocol-defined toxicity criteria, and all abnormal laboratory and vital signs findings that met grading criteria were considered AEs. For participants who enrolled under protocol v11.0, AEs were graded according to the NCI CTCAE, Version 5.0, and only clinically significant or related abnormal laboratory or vital signs findings were considered AEs.
Arm/Group | Cohort 1 - SAR440894 0.3 mg/kg | Cohort 2 - SAR440894 1 mg/kg | Cohort 3 - SAR440894 3 mg/kg | Cohort 4 - SAR440894 10 mg/kg | Cohort 5 - SAR440894 20 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 3/6 | 3/6 | 4/6 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - SAR440894 0.3 mg/kg (N=6) | Cohort 2 - SAR440894 1 mg/kg (N=6) | Cohort 3 - SAR440894 3 mg/kg (N=6) | Cohort 4 - SAR440894 10 mg/kg (N=6) | Cohort 5 - SAR440894 20 mg/kg (N=6) | Placebo (N=10)
Bradycardia (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (4) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 4 (17) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (11)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 3 (8) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (9) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (8)
Protein total decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cells urine positive (Investigations) | 2 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Respiratory rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT04441905/Prot_001.pdf
  • Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT04441905/SAP_002.pdf
  • Informed Consent Form (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT04441905/ICF_000.pdf